CLINICAL TRIAL: NCT05278858
Title: Needle-free Delivery of Intralesional Triamcinolone for Pediatric Alopecia Areata: a Pilot Study of Patient Tolerability
Brief Title: Needle-free Delivery of Intralesional Triamcinolone for Pediatric Alopecia Areata
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Lack of participants
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 20211626
Record Dates: First submitted 2022-01-26; First posted 2022-03-14 (Actual); Results first posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: Alopecia Areata
Keywords: Pediatric
MeSH Terms: conditions — Alopecia Areata

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- MedJet Device (Experimental): The Med-Jet-MBX needle-free injector (Med-Jet) is a novel, needle-free drug-delivery system, which we believe may be a solution to the pain and fear associated with needles. It uses regulated compressed air as a power source to accelerate an injectable fluid through a 0.005" orifice (6x smaller than a 30G needle) to penetrate the skin and deliver medication to a specific anatomical region (MedJet) The drug-delivery device is highly configurable allowing adjustable depth and volume parameters (MedJet). In addition, the high-performance design allows for triggering multiple injection sites rapidly which is practical when needing to treat large surface areas (MedJet).
  Interventions: Combination Product: MedJet Device with intralesional triamcinolone

INTERVENTIONS:
Combination Product: MedJet Device with intralesional triamcinolone — A standard sterile disposable 5 ml syringe will be used to draw TAC using standard sterile protocol. This syringe will be attached to the Med-Jet along with a sterile barrel and disposable sterile tip. The target lesion will be wiped with alcohol and injected with 10mg/ml of TAC directed towards the dermis to create a blanching wheal that is 1 cubic centimeter (total of 0.1 ml of injected fluid). The optimal injection pressure used on the subject will start at 110 pounds per square inch (psi) and increased by 10 psi until a blanching wheal is observed. The optimal pressure will be recorded. The injections will be repeated multiple times at the optimal pressure until the targeted patch is completely treated.

SUMMARY:
This is an interventional pilot study assessing the tolerability of needle-free delivery administration of ILTA with the Med-Jet as an alternative to conventional syringe and needle in patients with patchy pediatric alopecia areata. There will be a total of four (4) or five (5) visits necessary for study participation. The investigators hypothesize that the Med-Jet will have acceptable pain tolerability, efficacy, safety, and a positive impact on patient quality of life.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with alopecia areata by either:

  * A board-certified dermatologist, OR
  * Dermatology Nurse Practitioner, OR
  * Skin punch biopsy
* Patient has at least 2 alopecic patches each measuring at least 2 cm2 and are…

  * Located on contralateral body sites OR
  * Within the same body site but separated by ≥ 1 cm
* Patient is a candidate for intralesional triamcinolone.
* Patient able to give informed assent under IRB approval procedures when appropriate.
* At least one parent or guardian is able to provide informed consent.

Exclusion Criteria:

* Patient has alopecia totalis, alopecia universalis, or alopecia areata with ophiasis pattern.
* Known allergy or hypersensitivity to triamcinolone acetonide
* Pregnant, breastfeeding, or planning to get pregnant 4 weeks before, during, and 4 weeks after the study.
* Patient is unable/unwilling to provide informed assent when applicable.
* Known medical diagnosis or use of a medication that alters pain response at time of injection.
* Active infection at site designated for injection.
* If currently being treated for alopecia areata, the current treatment regimen has been started within less than 4 weeks of screening.

Ages: 6 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 3 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2023-06-06 (Actual); Study Completion 2023-06-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sonal Shah, MD, Principal Investigator — University Hospitals Cleveland Medical Center
Locations (1):
- University Hospitals Cleveland Medical Center, Cleveland, Ohio, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Recruited from UH derm providers who referred interested patients
Period: Overall Study
Arm/Group | MedJet Device
Started | 3
Completed | 2
Not Completed | 1
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | MedJet Device
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 0
  Unknown or Not Reported | 3
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 0
  More than one race | 0
  Unknown or Not Reported | 3

OUTCOME MEASURES:

1. Primary Outcome: Determine Patient Tolerability of Needle-free Delivery of Intralesional Triamcinolone Using the Patient-reported Outcomes of a Pain Score Assessment and a Patient Survey.
Description: For the pain score assessment, patients will rate their pain from the needle-free injection using the Wong-Baker FACES Scale and a numerical rating scale, in which score ranges from 0-10 where 0 is no pain and 10 is the worst pain imaginable.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 3
score on a scale | 3.7 (2.9)

2. Secondary Outcome: Change in Patient Reported Hair Loss
Description: The patient-reported efficacy assessments will consist of the Patient-Reported Hair Loss and the 5-Point Patient-Reported. The Patient-Reported Hair Loss assessment includes 5 categories to assess how much of the patient's scalp is missing hair. Reported on a scale of 0-4, with 0 being no hair loss, and 4 nearly all or all hair loss.
Time Frame: Baseline (pre-treatment), 12 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale
  Pre-treatment | 1.5 (0.5)
  Post-treatment | 1 (0)

3. Secondary Outcome: Patient Reported Hair Regrowth
Description: The 5-Point Patient-Reported Regrowth will ask the subject about their perceived amount of hair regrowth. Reported on a scale of 0-4, with 0 being no regrowth, and 4 being 100% regrowth.
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale | 2.5 (0.5)

4. Secondary Outcome: Change in Severity of Alopecia Tool (SALT) Score
Description: SALT Score is a score of 0-100, where 0 is no hair loss, and 100 is complete hair loss.
Time Frame: Baseline (Pre-treatment), 12 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale
  Pre-treatment | 28.8 (23.7)
  Post-treatment | 11.2 (11.2)

5. Secondary Outcome: Change in Alopecia Areata- Investigator Global Assessment (AA-IGA)
Description: AA-IGA is measured on a score of 1-5, with 1 being mild hair loss, to 5 being severe hair loss.
Time Frame: Baseline (Pre-treatment), 12 weeks (Post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale
  Pre-treatment | 3 (1)
  Post-treatment | 2 (1)

6. Secondary Outcome: Hair Regrowth of Treated Patch
Description: Scored on a 0-5 scale, with 5 being complete regrowth and 0 being further hair loss
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale | 4.5 (0.5)

7. Secondary Outcome: Hair Regrowth of Non-treated Patch
Description: Scored on a 0-5 scale, with 5 being complete regrowth and 0 being further hair loss
Time Frame: 12 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 2
score on a scale | 4.5 (0.5)

8. Secondary Outcome: Determine the Impact of Needle-free Delivery of Intralesional Triamcinolone on Quality of Life for Pediatric Alopecia Areata Using a Quality of Life Assessment.
Description: At each visit, subjects will answer either the Children's Dermatology Quality of Life Index (cCDLQI) (ages 6-11) or the Teenager's Quality of Life Index (T-QoL) (ages 12-17). Both the cCDLQI and T-QoL have the same scale ranges and directionality- 10 item questionnaire asking about skin troubles on a scale of 1-4, with 1 being "not at all" and 4 being "very much".
Time Frame: Baseline (pre-treatment), 12 weeks (post-treatment)
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | MedJet Device
Number analyzed (Participants) | 1
score on a scale
  Pre-treatment | 4 (3)
  Post-treatment | 2 (3.1)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | MedJet Device
All-Cause Mortality (participants affected / at risk) | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3
Other Adverse Events (participants affected / at risk) | 1/3
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MedJet Device (N=3)
Skin atrophy (Skin and subcutaneous tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2022-01-25): https://cdn.clinicaltrials.gov/large-docs/58/NCT05278858/Prot_SAP_000.pdf